CLINICAL TRIAL: NCT03175939
Title: Elimination of Adjuvant Chemotherapy for Selected Stage II and III Nasopharyngeal Carcinoma After Concomitant Radiotherapy And Chemotherapy
Brief Title: Elimination of Adjuvant Chemotherapy for Selected Stage II and III Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jia-Shing Wu, Attending Physician, M.D., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC9801
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Nasopharyngeal Cancer
Keywords: adjuvant chemotherapy; NPC
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Radiotherapy; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCRT alone (Experimental): External beam radiotherapy > 66 Gy Cisplatin 60 mg/m2 IV D1, 5-FU 600 mg/m2 IV D1-5 at week 1 and 5 of radiotherapy Modified for IMRT: Cisplatin 60 mg/m2 IV D1, 5-FU 600 mg/m2 IV D1-3 at week 1, 4 and 7 of radiotherapy
  Interventions: Radiation: Radiotherapy; Drug: Cisplatin; Drug: 5-FU

INTERVENTIONS:
Radiation: Radiotherapy — External beam radiotherapy with curative intent, at least 66 Gy
Drug: Cisplatin — cisplatin IV injection over 3 hours
  Other Names: CDDP
Drug: 5-FU — 5-FU IV 24 hours continuous infusion
  Other Names: 5-fluorouracil

SUMMARY:
This study evaluates whether some patients with nasopharyngeal carcinoma but with low risk of distant metastasis can be treated with only radiotherapy and concomitant chemotherapy but without additional adjuvant chemotherapy.

DETAILED DESCRIPTION:
The standard treatment for stage II-III nasopharyngeal carcinoma is radiotherapy with concomitant chemotherapy and adjuvant chemotherapy. A subset of these patients has very low risk for distant metastasis that adjuvant chemotherapy is probably unnecessary. The investigators would like to know if same therapeutic effect and survival rate can be achieved without adjuvant chemotherapy, (i.e. less chemotherapy, same effect)

ELIGIBILITY:
Inclusion Criteria:

* (1) biopsy-proven carcinoma of the nasopharynx,
* (2) AJCC 1997 Stage II (T2aN0, T1-T2aN1) or III (T1-T2aN2) disease,
* (3) normal renal function (Cr < 1.6 mg/dl),

Exclusion Criteria:

* open-neck lymph node biopsy
* previous chemotherapy or radiotherapy to the head and neck region
* distant metastasis or other malignant diseases except skin cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 1998-04-01 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Distant-metastasis-free survival | 5 years
  percentage of patients who survived and has no distant metastasis

SECONDARY OUTCOMES:
overall survival | 5 years
  percentage of patients who survived
disease-free survival | 5 years
  percentage of patients who survived and had no disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Skye Hung-Chun Cheng, M.D., Principal Investigator — Koo Foundation Sun Yat-Sen Cancer Center

IPD SHARING:
Plan to Share IPD: No